CLINICAL TRIAL: NCT00065117
Title: Safety, Tolerability and Efficacy of ZD6126 in Combination With Oxaliplatin, 5-Fluorouracil and Leucovorin in Subjects With Metastatic Colorectal Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2820C00007; 6126IL/00007
Record Dates: First submitted 2003-07-17; First posted 2003-07-18 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Colorectal Neoplasms; Metastases, Neoplasm
Keywords: metastatic; colorectal; first-line; adjuvant; cancer; Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — N-acetylcochinol-O-phosphate; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: ZD6126
Drug: Placebo
Drug: 5-fluorouracil
Drug: leucovorin
Drug: oxaliplatin

SUMMARY:
The purpose of this study is to assess the Safety, Tolerability and Efficacy of ZD6126 in Combination with Oxaliplatin, 5-Fluorouracil and Leucovorin in Subjects with Metastatic Colorectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal carcinoma
* Suitable for first-line treatment of metastatic disease

Exclusion Criteria:

* Peripheral neuropathy greater than Grade 1
* Adjuvant therapy within 6 months prior to study treatment
* Prior oxaliplatin
* Prior pelvic or whole abdomen radiation
* Any history of coronary angioplasty or history of myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2003-09; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Chicago, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Pittsburgh, Pennsylvania